CLINICAL TRIAL: NCT03021330
Title: Efficacy of Intermediate-Dose Cytarabine Induction Regimen in Adult AML
Status: Active, not recruiting | Phase: Phase 3 | Type: Interventional
Sponsor: Institute of Hematology & Blood Diseases Hospital, China (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: IIT2016007（Cytarabine）
Record Dates: First submitted 2017-01-12; First posted 2017-01-13 (Estimated); Last update posted 2025-05-30 (Actual); Status verified 2025-05

CONDITIONS: AML
MeSH Terms: interventions — Daunorubicin; Cytarabine

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- DA Regimen (Active Comparator): Patients receive standard DA induction regimen including daunomycin and cytarabine.
  Interventions: Drug: Daunomycin and Cytarabine (DA Regimen)
- Intermediate Dose of DA Regimen (Experimental): Patients receive DA induction regimen including daunomycin and intermediate dose of cytarabine.
  Interventions: Drug: Daunomycin and Cytarabine (Intermediate Dose of DA Regimen)

INTERVENTIONS:
Drug: Daunomycin and Cytarabine (DA Regimen) — Cytarabine at a dose of 100mg/㎡/d on day 1-7.
  Daunomycin at a dose of 60mg/㎡/d on day 1-3.
  Other Names: Daunomycin and Cytarabine
  Arms: DA Regimen
Drug: Daunomycin and Cytarabine (Intermediate Dose of DA Regimen) — Cytarabine at a dose of 100mg/㎡/d on day 1-4 and 1g/㎡/d on day 5-7.
  Daunomycin at a dose of 60mg/㎡/d on day 1-3.
  Other Names: Daunomycin and Cytarabine
  Arms: Intermediate Dose of DA Regimen

SUMMARY:
In this open-label, randomized, prospective clinical trial, newly-diagnosed AML patients will be randomized into 2 groups. In the experimental arm, patients receive DA induction regimen with intermediate dose of cytarabine. In the control arm, patients receive DA regimen with standard dose of cytarabine.The efficacy of induction therapy containing intermediate dose of cytarabine is evaluated and adverse events associated with treatment are recorded.The primary end point is overall survival.

DETAILED DESCRIPTION:
In this open-label, randomized, prospective clinical trial, newly-diagnosed AML patients will be randomized into 2 groups. In the experimental arm, patients receive DA induction regimen with intermediate dose of cytarabine at at a dose of 100mg/㎡/d on day 1-4 and 1g/㎡/Q12h on day5-7. In the control arm, patients receive DA regimen with standard dose of cytarabine at a dose of 100mg/㎡/d on day 1-7. Patients receive consolidation therapy containing high-dose cytarabine after achieved complete remission. Stem-cell transplantation is permitted for patients with intermediate- or poor-risk disease. The efficacy of induction therapy containing intermediate dose of cytarabine is evaluated and adverse events associated with treatment are recorded.The primary end point is overall survival.

ELIGIBILITY:
Inclusion Criteria:

1. Age of 14 to 55 years old;
2. Patients that meet the diagnostic criteria(WHO 2008 criteria) of AML (except APL subtypes).
3. ECOG score ≤ 2;
4. Patients with eligible laboratory examination including liver,renal and heart function.
5. Adult patients are willing to participate in the study and sign the informed consent by themselves or by their immediate family. Patients under 18 years old willing to participate should have their legal guardians sign the informed consent.

Exclusion Criteria:

1. Patients who had received induction therapy.
2. Secondary leukemia.
3. Patients had other tumor at active stage or had received radiotherapy or chemotherapy in the last 6 months due to other tumor.
4. Patients with other blood diseases(for example, haemophiliacs) are excluded.However, patients with abnormal blood count, but with undiagnosed MDS or MPD patients are included.
5. Acute panmyelosis with myelofibrosis and myeloid sarcoma patients;
6. With BCR-ABL fusion gene;
7. Pregnant or lactating women;
8. AML with ineligible renal or liver function;
9. AML with active cardiovascular disease;
10. Severe infection disease including uncured tuberculosis pulmonary aspergillosis;
11. AIDS;
12. Patients had central nervous system involvement when they were diagnosed as AML.
13. Patients with epilepsy or dementia or other mental disease who couldn't understand or follow the research.
14. Drugs, medical, mental or social situation may distract patients from following the research or being evaluated the results.
15. Patients with other factors which were considered unsuitable to participate in the study by the investigators.

Ages: 14 Years to 55 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult
Enrollment: 1100 (Estimated)
Dates: Start 2017-02-08 (Actual); Primary Completion 2026-05-15 (Estimated); Study Completion 2027-10-15 (Estimated)

PRIMARY OUTCOMES:
Overall Survival Rate (OS) | Within 5 years after randomization
  OS is defined as the time from the date of randomization until the date of death from any cause.

SECONDARY OUTCOMES:
Complete Remission Rate | Within 2 months after randomization
Event-Free Survival Rate | Within 5 years after randomization
Relapse-Free Survival Rate (RFS) | Within 5 years after randomization
Cumulative incidence of relapse | Within 5 years after randomization
Early Mortality | within 45 days after randomization

CONTACTS AND LOCATIONS:
Overall Officials: Jianxiang Wang, Dr, Principal Investigator — Institute of Hematology & Blood Diseases Hospital, China
Locations (1):
- Institute of Hematology & Blood Diseases Hospital, Tianjin, Tianjin Municipality, China

IPD SHARING:
Plan to Share IPD: No